CLINICAL TRIAL: NCT01731444
Title: Phenylephrine Tumescence for Hemostasis in Surgery for Burn Injury - A Randomized Control Trial
Brief Title: Phenylephrine Tumescence for Hemostasis in Surgery for Burn Injury
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PhenylephrineRCT
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Blood Loss, Surgical
Keywords: blood loss; burn; hemostasis
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage; Burns | interventions — Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phenylephrine (Experimental): 20 ug/cc
  Interventions: Drug: Phenylephrine
- Epinephrine (Active Comparator): 1:1000000
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Phenylephrine

SUMMARY:
The standard of care for treatment of burn injury is to inject a solution of epinephrine under the skin of the injured site in order to reduce blood loss during skin grafting. This solution of epinephrine has been shown to have effects on the body outside the donor site. Some people have increases in heart rate and blood pressure. We will study the effect of a phenylephrine solution in place of an epinephrine solution to control blood loss. We think that phenylephrine will help decrease blood loss and not change blood pressure or heart rate.

The injured area will be injected under the skin and a skin graft will be taken in the same way as we usually do. The only change will be the use of phenylephrine in the solution instead of epinephrine.

Our goal is to find whether or not phenylephrine or epinephrine solution results in a reduction of blood loss without affecting the rest of the body.

ELIGIBILITY:
Inclusion Criteria

a) Burn injury requiring debridement and grafting between 5-30% TBSA

Exclusion Criteria

1. Head and neck, hand, foot, or genital burns
2. On anticoagulants (except NSAIDs)
3. On monoamine oxidase inhibitor or tricyclic antidepressant
4. Coronary or peripheral vascular disease
5. History of arrhythmias
6. On a Beta-blocker
7. History of vascular abnormality
8. Hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mean arterial blood pressure (MAP) | during first 30 minutes
  Mean arterial blood pressure

SECONDARY OUTCOMES:
Blood Pressure | q15 min
  Cut off for safety: Diastolic >140 or Systolic >180;
  Recorded:
  * just prior to induction of anesthesia
  * maximum heart rate during time of procedure
  * minimum heart rate during time of procedure
Heart Rate | q15 min
  Recorded:
  * just prior to induction of anesthesia
  * maximum heart rate during time of procedure
  * minimum heart rate during time of procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada